CLINICAL TRIAL: NCT06696170
Title: Initial Safety and Performance of the CellFX® Nano-PFA 360 Catheter Endocardial Ablation System for the Treatment of Atrial Fibrillation
Brief Title: CellFX® Nanosecond Pulsed Field Ablation (PFA) 360 Catheter Ablation System for Treatment of Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-CCF-033
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation Paroxysmal; Cardiac Ablation; Cardiac Arrhythmia
Keywords: nsPFA; CellFX; Pulsed Field Ablation; nano-PFA
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CellFX nano-PFA Treatment Arm (Experimental): CellFX nano-PFA 360 Endocardial Ablation Catheter System
  Interventions: Device: CellFX nano-pFA 360 Endocardial Ablation Catheter System

INTERVENTIONS:
Device: CellFX nano-pFA 360 Endocardial Ablation Catheter System — The CellFX nano-PFA 360 Endocardial Ablation Catheter System includes the nano-pFA 360 Endocardial Ablation Catheter, CellFX Console, switcher box/adapter, and sensing cable. The System is a proprietary endocardial catheter system designed for use in cardiac electrophysiology procedures for the treatment of arrhythmias, including atrial fibrillation. The nano-PFA 360 Catheter ablates cardiac tissue using nonthermal nano-second pulses of electrical energy. Nanosecond Pulsed Field Ablation (nsPFA or nano-PFA) is a cell-specific, nonthermal ablation technology that delivers nanosecond-duration pulses of high-amplitude electrical energy to tissue via bipolar electrodes. The pulses disrupt the ability of the cell and internal organelles to maintain cellular homeostasis by creating nanopores in lipid membranes, ultimately leading to regulated cell death (RCD).

SUMMARY:
The objective of this study is to demonstrate initial safety and effectiveness of the CellFX nano-second Pulsed Field Ablation (nsPFA or nano-PFA) 360 Catheter Endocardial Ablation System in treating subjects with atrial fibrillation.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, open labelled, single-arm first-in-human (FIH) feasibility study to evaluate the initial clinical safety and device performance of the nano-PFA 360 Catheter Endocardial Ablation System for the treatment of atrial fibrillation. Enrolled subjects will be followed for up to 12 months post-nano PFA 360 Catheter Ablation. All subjects will undergo an electroanatomical mapping procedure post-ablation to evaluate immediate pulmonary vein isolation (PVI) and at 3 months post-index procedure to assess electrical isolation of the pulmonary veins.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 and ≤ 75 years of age on the day of enrollment
* Subject is willing and capable of providing Informed Consent to undergo study procedures and participate in all examinations and follow-up visits and tests associated with this clinical study
* Subjects with PAF who have had at least one AF episode documented within one (1) year prior to enrollment. Documentation may include ECG, transtelephonic monitor (TTM), Holter monitor (HM), or telemetry strip
* Subjects who have failed at least one antiarrhythmic drug (AAD; class I or III, or AV nodal blocking agents such as beta blockers and calcium channel blockers) as shown by recurrent symptomatic AF, or intolerance to the AAD or AV nodal blocking agents
* Antero-posterior left atrial diameter ≤ 5.5 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT) within 3 months prior to the procedure
* Left ventricular ejection fraction ≥ 40% as documented by TTE within 12 months prior to the procedure
* Received a standard cardiac work up and is an appropriate candidate for an investigational procedure as determined by the study investigators

Exclusion Criteria:

* Subject has an implantable electronic medical device. (i.e., pacemaker, ICD or CRT) or left atrial appendage device
* Subject has a prosthetic heart valve
* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* AF episodes lasting > 7 days
* Previous ablation for AF
* Subjects on amiodarone at any time during the past 3 months prior to enrollment
* Prior history of pericarditis or pericarditis within 3 months based on the TTE examination
* Prior history of rheumatic fever
* Prior history of medical procedure involving instrumentation of the left atrium (previous ablation, atrial septal defect (ASD) closure, left atrial appendage occlusion)
* History of severe chronic gastrointestinal problems involving the esophagus, stomach and/or untreated acid reflux
* History of abnormal bleeding and/or clotting disorder
* Contraindication to anticoagulation (i.e., Heparin, Dabigatran, Apixaban, Vitamin K Antagonists such as Warfarin)
* Active malignancy or history of treated cancer within 24 months of enrollment
* Clinically significant infection or sepsis on the day of index procedure with either fever, leukocytosis or requiring intravenous antibiotics
* History of stroke or TIA within prior 6 months, or any prior intracranial hemorrhage or permanent neurological deficit
* New York Heart Association (NYHA) class IIIb or IV congestive heart failure and/or any heart failure hospitalization within 3 months prior to enrollment
* Body mass index > 35 kg/m2
* Estimate glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 or has ever received hemodialysis
* History of untreated and serious hypotension, bradycardia or chronotropic incompetence
* Any of the following within 3 months of enrollment:

  1. Major surgery except for the index procedure
  2. Myocardial infarction
  3. Unstable angina
  4. Percutaneous coronary intervention
  5. Sudden cardiac death event
  6. Left atrial thrombus that has not resolved as shown by TEE or CT
* Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
* History of pulmonary hypertension with pulmonary systolic artery pressure >50 mm Hg, severe Chronic Obstructive Pulmonary Disease or restrictive lung disease
* Subjects with any other significant uncontrolled or unstable medical condition (such as uncontrolled brady-arrhythmias, ventricular arrhythmias, hyperthyroidism or significant coagulation disorder)
* Life expectancy less than one year
* Clinically significant psychological condition that in the physician's opinion would prohibit the subject's ability to meet the protocol requirements.
* Females of childbearing potential who are nursing, pregnant, or planning to become pregnant during the study period
* Other criteria, which the Investigator determines would make the patient unsuitable to participate (e.g. uncontrolled drug and/or alcohol addiction, congenital disease, fragility)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
Rate of primary safety major adverse events (MAEs) | Within 30 days post-ablation procedure
  The primary safety endpoint includes major adverse events (MAEs) specifically related to the device or ablation procedure for the following
  * Asymptomatic Cerebral Embolism
  * Arterioesophageal Fistula
  * Bleeding Requiring Transfusion
  * Cardiac Perforation/Tamponade
  * Death
  * Esophageal Injury Resulting in Perforation
  * Myocardial Infarction
  * Pericarditis Requiring Intervention or Hospitalization
  * Phrenic Nerve Injury/Diaphragmatic Paralysis
  * Pulmonary Edema/Respiratory Insufficiency
  * Pulmonary Vein Stenosis (≥70% diameter reduction)
  * Stroke or Transient Ischemic Attack
  * Vagal Nerve Injury Resulting in Esophageal Dysmotility or Gastroparesis
  * Vascular Access Complication Requiring Intervention
Proportion of participants achieving acute procedural success. | Immediately post-ablation procedure
  Acute procedural success is achieving entrance block of the pulmonary veins

SECONDARY OUTCOMES:
Proportion of participants reporting one or more significant adverse events (SAEs) | Within 12 months post-ablation procedure
  Safety related to the reporting one or more SAEs for each follow-up interval as described.
  * Atrio-esophageal fistula (up to 3-month visit)
  * Pulmonary Vein (PV) stenosis (up to 3-month visit)
  * Subjects presenting with Primary SAEs up to the 12-month post- procedure follow-up
  * Subjects presenting with any AEs or SAEs up to the 12-month post- procedure follow-up
Proportion of participants achieving long-term technical success | Within 3 months post-ablation procedure
  Long-term technical success is defined as electrical isolation of the pulmonary veins (PVI) assessed during an electroanatomical mapping procedure.
Proportion of participants achieving treatment success | Within 12 months post-ablation procedure
  Treatment success is defined by freedom from the following failures:
  1. Recurrence of atrial fibrillation, atrial flutter, atrial tachycardia (AF/AFL/AT) as evidenced by episodes ≥ 30 secs on transtelephonic monitoring (TTM), Holter monitoring, or continuously 12-lead electrocardiogram (ECG)
  2. Cardioversion for atrial fibrillation (AF) /atrial flutter (AFL) / atrial tachycardia (AT)
  3. Repeat ablation failure
  4. Antiarrhythmic Drugs (AADs) failure
  5. Surgical treatment for AF/AFL/AT after the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Rich A. Nuccitelli, PhD, Study Director — Pulse Biosciences, Inc.
Locations (3):
- Hartcentrum Hasselt Research Center /Jessa Hospital, Hasselt, Belgium
- Na Homolce Hospital, Prague, Czechia
- Policlinico Tor Vergata Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No